CLINICAL TRIAL: NCT03914248
Title: Monitoring Large Vessel Vasculitis With PET/MR Imaging: an Exploratory Study
Brief Title: Monitoring Large Vessel Vasculitis With PET/MR Imaging
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: E182026
Record Dates: First submitted 2019-04-02; First posted 2019-04-16 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Large Vessel Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active large vessel vasculitis: PET/MR scan

SUMMARY:
Large vessel vasculitis (LVV) causes blood vessel inflammation leading to pain, fatigue and complications such as aneurysm formation and stroke. Treatments used can have significant side-effects. Doctors find it difficult to determine when to start and stop treatment, often leading to over- or under-treatment. A new test is required to determine disease activity that will guide treatment more accurately. This study will recruit participants with active LVV from throughout Scotland in order to assess the ability of two new types of scan - positron emission tomography with magnetic resonance imaging (PET/MR) and retinal optical coherence tomography (OCT) - to determine disease activity. In addition, I will investigate the link between LVV and heart disease.

DETAILED DESCRIPTION:
Large vessel vasculitis (LVV) is a multi-system, autoimmune disease characterised by non-specific symptoms, pain and high glucocorticoid requirements. The lack of a robust biomarker that tracks disease activity makes disease monitoring difficult. This leads to both disease over-treatment, resulting in adverse effects of glucocorticoids, and under-treatment, with the potential for significant vascular complications. Additionally, the link between LVV and cardiovascular disease (CVD), which is the main cause of death in these patients, remains poorly characterised. An imaging tool which is capable of accurately monitoring disease activity over time is urgently required. Positron emission tomography with magnetic resonance imaging (PET/MR) and retinal optical coherence tomography (OCT) have the potential to meet this need. PET/MR is uniquely useful for imaging CVD and utilises ~50% of the radiation dose of PET with computerised tomography. OCT is a novel potential biomarker of microvascular dysfunction, systemic inflammation and CVD risk in small vessel vasculitis. Participants with a new diagnosis or recent flare of LVV will undergo serial PET/MR and OCT scanning alongside established measures of CVD risk. Results will be compared with current clinical measures of disease activity and with banked control data.

ELIGIBILITY:
Inclusion Criteria:

* A new diagnosis of LVV or a known diagnosis of LVV presenting with disease relapse

Exclusion Criteria:

* Predominantly cranial symptoms
* LVV secondary to other conditions
* Treatment with high dose glucocorticoids for >2 weeks at time of recruitment
* Contraindication to MR or PET
* Unable to travel to Edinburgh
* Estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2
* Unable to provide informed consent
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from outpatient clinics throughout Scotland
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Maximum standardised uptake values (SUVmax) | 0 and 6 months
  Maximum standardised uptake values (SUVmax) will be assessed using PETMR. This information will be used to quantify disease activity and atheroma at pre-specified vascular segments.

SECONDARY OUTCOMES:
Choroidal thickness in microns | 0 and 6 months
  Assessment of choroidal thickness as measured using optical coherence tomography will be made at baseline and 6 months
Choroidal volume in mm3 | 0 and 6 months
  Assessment of choroidal volume using optical coherence tomography will be made at baseline and 6 months
Retinal vasculature morphology | 0 and 6 months
  Visual assessment of arteriolar thickness, branching coefficient and branching angle, fractal dimension, and venular tortuosity will be made using OPTOS imaging at baseline and 6 months
24-hour ambulatory blood pressure in mmHg | 0 and 6 months
  Assessment of 24-hour ambulatory systolic and diastolic blood pressure will be made at baseline and 6 months
Pulse wave velocity | 0 and 6 months
  Assessment of arterial stiffness will be made using pulse wave velocity as measured using SphygmoCor technology. Percentage change in pulse wave velocity will be compared between baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MBChB PhD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided